CLINICAL TRIAL: NCT05399524
Title: FUTURE-GB Trial (Functional and Ultrasound-guided Resection of Glioblastoma) A 2-Stage Trial. A Learning Phase Evaluation of Participating Centres, Followed by a Randomised, Controlled Multicentre Phase III Trial.
Brief Title: Functional and Ultrasound Guided Resection of Glioblastoma
Acronym: FUTURE-GB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other); Efficacy and Mechanism Evaluation (EME) Programme (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14763
Record Dates: First submitted 2021-11-24; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-04

CONDITIONS: Glioma Glioblastoma Multiforme
Keywords: DTI; iUS
MeSH Terms: conditions — Glioblastoma | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: FUTURE-GB is a 2-Stage trial: Stage 1 is a non-randomised multicentre learning and evaluation Stage (IDEAL IIB study), and Stage 2 a prospective, multicentre definitive randomised controlled trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Additional pre- and intra-operative imaging (Experimental): Surgery to resect the GB using Diffusion Tensor Imaging (DTI) and intraoperative Ultrasound (iUS) (navigated iUS where available) in addition to standard care (i.e. neuronavigation based on preoperative MRI and intraoperative use of 5-aminolevulinic acid (5-ALA))
  Interventions: Other: Additional pre- and intra-operative imaging
- Standard of Care (Active Comparator): The comparator is standard care as per current NICE guidelines (i.e. neuronavigation based on preoperative MRI and intraoperative use of 5-ALA).
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Standard of Care — Neuronavigation and intraoperative 5-ALA
  Arms: Standard of Care
Other: Additional pre- and intra-operative imaging — Additional DTI scan during routine pre-operative tumour MRI scan, additional use of intraoperative ultrasound in addition to normal to standard of care (Neuronavigation and intraoperative 5-ALA)
  Other Names: DTI; IUS
  Arms: Additional pre- and intra-operative imaging

SUMMARY:
Functional and ultrasound-guided resection of glioblastoma: assessing the use of additional imaging during surgery to improve outcomes for patients with glioblastoma brain tumours

DETAILED DESCRIPTION:
Stage 1 (IDEAL IIB study) of the trial is observational only and all participants will receive all technologies during surgery.

Stage 2 will be randomised. Randomisation will be via the web-based service provided by the Oxford Clinical Trials Research Unit (OCTRU), using the method of minimisation. Participants will be randomised 1:1 to either:

1. Standard care surgery (neuronavigation based on preoperative imaging and intraoperative use of 5-ALA)(Control arm)
2. Standard care surgery (neuronavigation based on preoperative imaging and intraoperative use of 5-ALA) AND of DTI neuronavigation and NiUS (Intervention arm)

At baseline all participants will undergo a routine preoperative neuronavigation MRI scan. Those participants randomised to the experimental arm, will also have a DTI scan (additional 5 minutes in the MRI). All participants will then undergo the planned resection of their tumour, with the additional technologies if they are in the experimental arm. Following surgery, participants in both arms have the same follow up schedule and undergo standard clinical care for a total of 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Neuro-oncology Multi-Disciplinary Team (MDT) decision that the imaging shows a primary GB tumour which is maximally resectable (attempted gross total resection of all enhancing tumour)
* Patient is suitable for concomitant adjuvant radiotherapy and Temozolomide (TMZ) chemotherapy or adjuvant TMZ at the time of MDT decision
* Able to receive 5-ALA
* Willing and able to give informed consent
* Able to complete trial questionnaires, this may be with support where English is not their first language. (Stage 2 only)
* Able to provide a proxy who is willing to complete questionnaires as requested (Stage 2 only).

Exclusion Criteria:

* Midline/basal ganglia/cerebellum/brainstem GB
* Multifocal GB
* Recurrent GB
* Suspected secondary GB
* Contraindication to MRI

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Stage 1 Primary Outcome: to demonstrate the feasibility of using DTI and iUS in addition to standard of care for neurosurgery using a combination of qualitative and quantitative data to prove workflow capability at each site. | Measured 6 weeks post-surgery
  Sites are qualitatively assessed through a standardisation stage, providing feedback to enable learning and ensure the workflow is followed. Sites with satisfactory data will "progress" and pass into Stage 2.
  The measures assessed in combination are:
  1. Operation length, in normal range for this surgery.
  2. Use of DTI neuronavigation & iUS to achieve maximal safe tumour resection without major neurological deficit, measured by getting clear, relevant images for the DTI & US scans, and accurate pre-operative tractography.
  3. Extent of tumour resection (cm³ remaining) on postoperative MRI scan.
  4. Surgical Complications/Serious Adverse Events-measured from recorded post-operative complications and a 6-month notes check to ensure patient safety.
  If the assessment panel is satisfied with the data after ~3 recruits, a site will progress into Stage 2 of the trial, the RCT. Data will be analysed for Stage 1 once all sites have progressed through into Stage 2 of the trial.
Stage 2 Primary Outcome: to assess whether additional imaging to standard of care changes Deterioration Free Survival (DFS) (Where deterioration relates to global health status only) | Measured from baseline up to 24 months
  This is measured by a composite of:
  1. Change in global health status domain of the QLQ-C30 questionnaire (Quality of Life Questionnaire Cancer) from baseline to final questionnaire completion. Questionnaires are administered at baseline, 6 weeks, then every 3 months until 24months.
  2. Progression Free Survival (PFS). This is measured by radiological tumour progression on imaging, which is taken 3-months post-op and 3-monthly thereafter.
  3. Overall Survival (OS) with an event defined as either deterioration, progression or death.

SECONDARY OUTCOMES:
Stage 2: To assess if additional intraoperative imaging changes DFS where deterioration relates to physical and social functioning, and motor and communication dysfunction | Measured from baseline up to 24 months
  This is measured using a combination of specific questions (physical functioning and social functioning) in the QLQ-C30 (Quality of Life Questionnaire Cancer) and BN20 questionnaire (Quality of Life Questionnaire Brain) (motor dysfunction and communication deficit questions), combined with the values of Progression Free Survival (PFS) and overall survival (OS) taken from the primary outcome.
  Questionnaires are administered at baseline, 6 weeks, then every 3 months until 24months.
Stage 2: To assess whether additional intraoperative imaging to standard of care changes time to deterioration | Measured from baseline up to 24 months
  Defined similar to DFS with the exception that progression is excluded as an event (i.e. only deterioration or death are considered). There will be five time to deterioration outcomes, one for each of the domains utilised in the primary and secondary DFS outcomes, used in turn to define deterioration
Stage 2: To assess whether additional intraoperative imaging to standard of care improves Overall Survival (OS) | To be recorded at 24 months
  OS (time from randomisation to death or trial closure)
Stage 2: To assess whether additional intraoperative imaging (DTI and iUS*) to standard of care (Neuronavigation and intraoperative 5-ALA) changes Progression Free Survival (PFS) | MRI at 6 months post-op., and then 3 monthly up to 24 months or an MRI performed outside protocol if patient is symptomatic
  PFS (time from randomisation to radiological tumour progression on imaging, as agreed in local MDT
  This involves using the post-operative MRI scan as a reference point and making comparisons will the ensuing MRI reports that are recieved 3 months post-surgery and 3 monthly thereafter until 24 months post-surgery.
Stage 2: To assess whether additional intraoperative imaging (DTI and iUS*) to standard of care (Neuronavigation and intraoperative 5-ALA) changes the extent of tumour resection | Measured 1 week post-surgery
  Extent of resection as percent of pre-operative tumour volume on postoperative contrast enhanced MRI
Stage 2: To assess whether additional intraoperative imaging (DTI and iUS*) to standard of care (Neuronavigation and intraoperative 5-ALA) changes the incidence of surgical complications | Measured from surgery up to 24 months
  Number and type of surgical complications
Stage 2: To assess whether additional intraoperative imaging (DTI and iUS*) to standard of care (Neuronavigation and intraoperative 5-ALA) changes the number of patients eligible for adjuvant treatment following surgery | Measured 3 months post surgery
  Number of patients eligible for adjuvant treatment
Stage 2: To assess whether additional intraoperative imaging (DTI and iUS*) to standard of care (Neuronavigation and intraoperative 5-ALA) changes functional outcome postoperatively | Measured from baseline up to 24 months
  Measured by any change in the functional performance assessment which consistes of a combination of:
  1. The WHO (World Health Organisation) performance status
  2. A 5-minute telephone mini-MoCA (The Montreal Cognitive Assessment, Montreal Version)
  3. Barthel Index
  4. MRC (Medical Research Council) grading of power in all 4 limbs
  Assessments are made at baseline, at hospital discharge, 6 weeks post-op, 3 months post-op, then 3 monthly thereafter until 24 months.
Stage 2: Assess the correlation of proxy to participant classification assessment of quality of life | Measured from baseline up to 24 months. Proxy will not complete questionnaires when participant stops completing them.
  Assessed using comparisons between the patient and proxy responses to the Quality of Life questionnaires administered. Specifically comparisons between the answers to questions 29 and 30 of the QLQ-C30.

OTHER OUTCOMES:
Tertiary Mechanistic Objectives (on a sub set of participants): assessment of the sensitivity and specificity of the anatomico-spatial location of DTI fibre tracts compared to Standard of Care | 6 weeks post-surgery
  To assess the sensitivity and specificity of the anatomico-spatial location of DTI fibre tracts compared with intraoperative direct electrical stimulation/behavioural change without stimulation but related to adjacent white fibre tract in patients undergoing awake surgery, or motor evoked potential changes in patients undergoing surgery.
  Measured by sensitivity and specificity calculation using pre and post-surgery MRI images
Tertiary Mechanistic Objectives (on a sub set of participants): assessment of the sensitivity and specificity of iUS to identify the tumour boundary when compared with 5-ALA. | 6 weeks post-surgery
  To assess the sensitivity and specificity of iUS* to identify the tumour boundary when compared with 5-ALA, navigated biopsies will be taken from tumour boundary tissue planned for resection.
  Intra operative iUS* images and post-operative MRI scans and Intraoperative biopsy samples

CONTACTS AND LOCATIONS:
Overall Officials: Puneet Plaha, Study Director — University of Oxford
Locations (24):
- United Kingdom (24):
  - Queen Elizabeth Hospital, University Hospitals Birmingham NHSFT, Birmingham
  - Royal Sussex County Hospital, Brighton
  - Southmead Hospital, North Bristol NHST, Bristol
  - Addenbrookes Hospital, Cambridge University NHSFT, Cambridge
  - University Hospital of Wales, Cardiff & Vale University Health Board, Cardiff
  - University Hospital, Coventry, Coventry
  - Ninewells Hospital, NHS Tayside, Dundee
  - The Royal Infirmary of Edinburgh, NHS Lothian, Edinburgh
  - Hull Royal Infirmary, Hull
  - Leeds General Infirmary, Leeds
  - The Walton Centre, Liverpool
  - Royal London Hospital, Barts Health NHS Trust, London
  - King's College Hospital, London
  - Charing Cross Hospital/St Mary's, Imperial College Healthcare NHS Trust, London
  - James Cook University Hospital, South Tees Hospitals NHSFT, Middlesbrough
  - Royal Victoria Infirmary, Newcastle upon Tyne Hospitals NHSFT, Newcastle upon Tyne
  - Queen's Medical Centre, Nottingham University Hospitals NHST, Nottingham
  - The John Radcliffe Hospital, Oxford University Hospitals NHSFT, Oxford
  - Derriford Hospital, University Hospitals Plymouth NHS Trust, Plymouth
  - Royal Preston Hospital, Lancashire Teaching Hospitals NHSFT, Preston
  - Queen's Hospital, Barking, Havering and Redbridge University Hospitals NHST, Romford
  - Royal Hallamshire Hospital, Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - Southampton General Hospital, University Hospital Southampton NHSFT, Southampton
  - Royal Stoke University Hospital, University Hospitals of North Midlands NHST, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/24/NCT05399524/Prot_000.pdf